CLINICAL TRIAL: NCT01369420
Title: A Safety Evaluation of the NanoKnife Low Energy Direct Current (LEDC) System in Subjects With Locally Advanced Unresectable Pancreatic Cancer - A Pilot Study
Brief Title: NanoKnife Low Energy Direct Current (LEDC) System in Subjects With Locally Advanced Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-208
Record Dates: First submitted 2011-06-07; First posted 2011-06-09 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: locoregional cancer therapy; pancreatic cancer; unresectable pancreatic cancer; pancreatic adenocarcinoma; locally advanced, unresectable pancreatic cancer; pancreatic cancer tumor ablation; NanoKnife tumor ablation for pancreatic cancer; NanoKnife LEDC system tumor ablation; Non thermal ablation; Irreversible electroporation for pancreatic cancer treatment; IRE for unresectable pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NanoKnife Low Energy Direct Current (LEDC) System Ablation — 90 pulses of 70 microseconds each in duration will be administered per electrode pair.
  Other Names: ◦ Low Energy Direct Current (LEDC) System; ◦ HVP01 Electroporation System; ◦ NanoKnife LEDC System; ◦ NanoKnife IRE System; ◦ Non-Thermal Irreversible Eletroporation (NTIRE) System; ◦ Angiodynamics IRE System; ◦ Non-Thermal Ablation

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of the NanoKnife Low Energy Direct Current (LEDC) System when used to treat unresectable pancreatic adenocarcinoma. Safety will be reviewed by means of analysis of adverse events, including serious adverse events, laboratory data, physician exam findings, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

1. male or female
2. >/= 18 years of age
3. meets criteria for locally advanced unresectable pancreatic adenocarcinoma, as radiographically proven pancreatic cancer as determined by a surgical oncologist via pancreatic CT or who were initially thought to be resectable; however at the time of surgery were upstaged to unresectability, via direct visualization
4. tumor size must be < 4 cm and must be measurable
5. must have an INR <1.5
6. must be unresponsive to chemotherapy as demonstrated with either CT or MR imaging and not have taken any chemotherapy agents within 14 days of treatment with the NanoKnife LEDC System
7. are willing and able to comply with the protocol requirements
8. are able to comprehend and willing to sign an Informed Consent Form (ICF)

Exclusion Criteria:

1. a baseline creatinine reported as > 2.0 mg/dL
2. have any reported baseline lab values with a grade 3 or 4 toxicity as defined by the CTCAE Version 3.0
3. inability to stop antiplatelet and Coumadin therapy for 7 days prior to and 7 days post treatment with the NanoKnife System
4. known history of contrast allergy that cannot be medically managed
5. known hypersensitivity to the metal in the electrodes (stainless steel 304L) that cannot be medically managed
6. unable to be treated with a muscle blockade agent (e.g. pancuronium bromide, atracurium, cisatracurium, etc)
7. women who are pregnant or currently breast feeding
8. women of childbearing potential who are not utilizing an acceptable method of contraception
9. have taken an investigational agent within 30 days of visit 1
10. have implanted cardiac pacemakers or defibrillators
11. have implanted electronic devices or implants with metal parts in the immediate vicinity of a lesion
12. have a history of epilepsy or cardiac arrhythmia (atrial or ventricular fibrillation)
13. have a recent history of myocardial infarction (within the past 2 months)
14. have Q-T intervals greater than 550 ms unless treated with an Accysync Model 72 synchronization system controlling the NanoKnife system's output pulses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety | 90 days
  * reported adverse events and adverse effects/events (serious and non serious),
  * unanticipated adverse events and device complaints,
  * safety laboratory tests (hematology, chemistry, amylase, lipase),
  * vital signs,
  * physical findings (including symptoms, vital signs and weight changes)

SECONDARY OUTCOMES:
Efficacy | 90 days
  Evaluation of short term efficacy based upon tumor evaluation and symptomatic response as defined by:
  * imaging will be used to evaluate changes in tumor size in addition to evaluating the completeness of ablation,
  * tumor evaluation by evaluating changes in CA-19-9 marker,
  * symptomatic changes of quality of life questionnaires,
  * physician assessment of the performance status of the subject,
  * pain assessment and subject analgesic consumption,
  * assessment of tumor for downstaging to resectability at the time of imaging

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Bassi, M.D., Principal Investigator — Policlinico "G.B. Rossi", University of Verona, Department of Surgery
Locations (1):
- Policlinico "G.B. Rossi", University of Verona, Department of Surgery, Verona, Verona, Italy

REFERENCES:
- [Background] Varshney S, Sewkani A, Sharma S, Kapoor S, Naik S, Sharma A, Patel K. Radiofrequency ablation of unresectable pancreatic carcinoma: feasibility, efficacy and safety. JOP. 2006 Jan 11;7(1):74-8. PMID 16407624
- [Background] Spiliotis JD, Datsis AC, Michalopoulos NV, Kekelos SP, Vaxevanidou A, Rogdakis AG, Christopoulou AN. Radiofrequency ablation combined with palliative surgery may prolong survival of patients with advanced cancer of the pancreas. Langenbecks Arch Surg. 2007 Jan;392(1):55-60. doi: 10.1007/s00423-006-0098-5. Epub 2006 Nov 7. PMID 17089173
- [Background] Hadjicostas P, Malakounides N, Varianos C, Kitiris E, Lerni F, Symeonides P. Radiofrequency ablation in pancreatic cancer. HPB (Oxford). 2006;8(1):61-4. doi: 10.1080/13651820500466673. PMID 18333241
- [Background] Wu Y, Tang Z, Fang H, Gao S, Chen J, Wang Y, Yan H. High operative risk of cool-tip radiofrequency ablation for unresectable pancreatic head cancer. J Surg Oncol. 2006 Oct 1;94(5):392-5. doi: 10.1002/jso.20580. PMID 16967436
- [Background] Matsui Y, Nakagawa A, Kamiyama Y, Yamamoto K, Kubo N, Nakase Y. Selective thermocoagulation of unresectable pancreatic cancers by using radiofrequency capacitive heating. Pancreas. 2000 Jan;20(1):14-20. doi: 10.1097/00006676-200001000-00002. PMID 10630378
- [Background] Elias D, Baton O, Sideris L, Lasser P, Pocard M. Necrotizing pancreatitis after radiofrequency destruction of pancreatic tumours. Eur J Surg Oncol. 2004 Feb;30(1):85-7. doi: 10.1016/j.ejso.2003.10.013. PMID 14736529
- [Background] Connor S, Raraty MG, Neoptolemos JP, Layer P, Runzi M, Steinberg WM, Barkin JS, Bradley EL 3rd, Dimagno E. Does infected pancreatic necrosis require immediate or emergency debridement? Pancreas. 2006 Aug;33(2):128-34. doi: 10.1097/01.mpa.0000234074.76501.a6. No abstract available. PMID 16868477
- [Background] Raraty MG, Connor S, Criddle DN, Sutton R, Neoptolemos JP. Acute pancreatitis and organ failure: pathophysiology, natural history, and management strategies. Curr Gastroenterol Rep. 2004 Apr;6(2):99-103. doi: 10.1007/s11894-004-0035-0. PMID 15191686
- [Background] Chan YC, Leung PS. Acute pancreatitis: animal models and recent advances in basic research. Pancreas. 2007 Jan;34(1):1-14. doi: 10.1097/01.mpa.0000246658.38375.04. PMID 17198179
- [Background] Freitag M, Standl TG, Kleinhans H, Gottschalk A, Mann O, Rempf C, Bachmann K, Gocht A, Petri S, Izbicki JR, Strate T. Improvement of impaired microcirculation and tissue oxygenation by hemodilution with hydroxyethyl starch plus cell-free hemoglobin in acute porcine pancreatitis. Pancreatology. 2006;6(3):232-9. doi: 10.1159/000091962. Epub 2006 Mar 9. PMID 16534248